CLINICAL TRIAL: NCT05479981
Title: A Phase 2 Extension Study to Evaluate the Long-Term Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of AOC 1001 Administered Intravenously to Adult Myotonic Dystrophy Type 1 (DM1) Patients
Brief Title: Extension of AOC 1001-CS1 (MARINA) Study in Adult Myotonic Dystrophy Type 1 (DM1) Patients
Acronym: MARINA-OLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avidity Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOC 1001-CS2
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: DM1; Muscular Dystrophies; Myotonic Dystrophy; Myotonic Dystrophy 1; Myotonic Disorders; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases
Keywords: DM1; Myotonic Dystrophy 1; Myotonic Dystrophy Type 1 (DM1); Myotonic Dystrophy; DM; Dystrophy Myotonic; Myotonic Disorders; Steinert Disease; MARINA-OLE; MARINA; Avidity Biosciences; Avidity; AOC 1001; Myotonic Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophies; Myotonic Dystrophy; Myotonic Disorders; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Masking Description: Participants will receive one blinded treatment at Day 43. Treatment assignment on this day will be based on treatment received in AOC 1001-CS1 so that participants who did not receive active drug on Day 43 in AOC 1001-CS1 will received active drug on Day 43 in AOC 1001-CS2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AOC 1001 (Experimental): AOC 1001 will initially be administered quarterly. On Day 43 patients will receive an additional dose. Treatment assignment will be based on treatment received in AOC 1001-CS1. If participant did not receive AOC 1001 on Day 43 in AOC 1001-CS1, participant will receive AOC 1001 treatment on Day 43 in AOC 1001-CS2. Beginning in September 2024, AOC 1001 will be administered every 8 weeks.
  Interventions: Drug: AOC 1001
- AOC 1001 (with Placebo at Day 43) (Experimental): AOC 1001 will initially be administered quarterly. On Day 43 patients will receive an additional dose. Treatment assignment will be based on treatment received in AOC 1001-CS1. If participant received AOC 1001 on Day 43 in AOC 1001-CS1, participant will receive blinded placebo treatment on Day 43 in AOC 1001-CS2. Beginning in September 2024, AOC 1001 will be administered every 8 weeks.
  Interventions: Drug: Placebo; Drug: AOC 1001

INTERVENTIONS:
Drug: Placebo — Placebo will be administered by intravenous (IV) infusion.
  Other Names: Saline
  Arms: AOC 1001 (with Placebo at Day 43)
Drug: AOC 1001 — AOC 1001 will be administered by intravenous (IV) infusion.

SUMMARY:
AOC 1001-CS2 (MARINA-OLE) is a Phase 2 extension of the AOC 1001-CS1 (MARINA) study to evaluate the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of multiple-doses of AOC 1001 Administered Intravenously to Adult Myotonic Dystrophy Type 1 (DM1) patients

DETAILED DESCRIPTION:
This study will continue to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of AOC 1001 in participants that enrolled in the randomized, placebo-controlled, First-In-Human Phase 1/2 AOC 1001-CS1 (MARINA) clinical study.

Participants from AOC 1001-CS1 are eligible to enroll in AOC 1001-CS2 if they have satisfactorily completed AOC 1001-CS1.

After completion of Q8W Visit 6 assessments, participants will have the option to enroll in another AOC 1001 open-label extension (OLE) study. Participants who do not enroll in an AOC 1001 OLE study will be monitored for safety for a total of 8 weeks from the last dose of study drug. Total duration on study is up to 37 months (3 years 1 month).

As of September 2024, the dosing regimen was updated to every 8 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Completion of AOC 1001-CS1 (MARINA) study with satisfactory compliance and no significant tolerability issues

Key Exclusion Criteria:

* Pregnancy, intent to become pregnant, or active breastfeeding
* Unwilling or unable to continue to comply with contraceptive requirements
* Any new conditions or worsening of existing conditions that in the opinion of the investigator or sponsor would make the participant unsuitable for the study or could interfere with participation or completion of the study

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Number and severity of treatment-emergent adverse events (TEAEs) | Through study completion

SECONDARY OUTCOMES:
AOC 1001 levels in muscle tissue | Through Day 183
Change and percentage change from baseline in DMPK mRNA knockdown | Through Day 183
Change and percentage change from baseline in Spliceopathy | Through Day 183
Plasma pharmacokinetic (PK) parameters | Up to Day 729
  Maximum and trough plasma concentration

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia